CLINICAL TRIAL: NCT05129423
Title: A Phase II, Multicenter, Randomized, Double-Blind, Placebo-Controlled Pilot and Dose-Ranging Study of MTPS9579A in Participants With Refractory Chronic Spontaneous Urticaria
Brief Title: A Study of MTPS9579A in Participants With Refractory Chronic Spontaneous Urticaria
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Development of MTPS9579A was terminated for strategic/business reasons.
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GA43512
Record Dates: First submitted 2021-11-05; First posted 2021-11-22 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Chronic Spontaneous Urticaria
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part 1: MTPS9579A Dose A (Experimental): In Part 1, participants will receive MTPS9579A dose A every 4 weeks from randomization to Week 12.
  Interventions: Drug: MTPS9579A
- Part 1: Placebo (Placebo Comparator): In Part 1, participants will receive placebo matched with MTPS9579A, every 4 weeks from randomization through Week 12.
  Interventions: Drug: Placebo
- Part 2: MTPS9579A Dose A (Experimental): In Part 2, participants will receive MTPS9579A dose A, every 4 weeks from randomization to Week 12.
  Interventions: Drug: MTPS9579A
- Part 2: MTPS9579A Dose B (Experimental): In Part 2, participants will receive MTPS9579A dose B, every 4 weeks from randomization to Week 12.
  Interventions: Drug: MTPS9579A
- Part 2: MTPS9579A Dose C (Experimental): In Part 2, participants will receive MTPS9579A dose C, every 4 weeks from randomization to Week 12.
  Interventions: Drug: MTPS9579A
- Part 2: MTPS9579A Dose D (Experimental): In Part 2, participants will receive MTPS9579A dose D, every 4 weeks from randomization to Week 12.
  Interventions: Drug: MTPS9579A
- Part 2: Placebo Dose A (Placebo Comparator): In Part 2, participants will receive placebo matched with MTPS9579A dose A and B, every 4 weeks from randomization through Week 12.
  Interventions: Drug: Placebo
- Part 2: Placebo Dose B (Placebo Comparator): In Part 2, participants will receive placebo matched with MTPS9579A dose C and D, every 4 weeks from randomization through Week 12.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MTPS9579A — MTPS9579A will be administered.
  Arms: Part 1: MTPS9579A Dose A; Part 2: MTPS9579A Dose A; Part 2: MTPS9579A Dose B; Part 2: MTPS9579A Dose C; Part 2: MTPS9579A Dose D
Drug: Placebo — Placebo matched with MTPS9579A will be administered.
  Arms: Part 1: Placebo; Part 2: Placebo Dose A; Part 2: Placebo Dose B

SUMMARY:
This pilot and dose-ranging study will evaluate the efficacy, safety, and pharmacokinetics of MTPS9579A compared with placebo in participants with chronic spontaneous urticaria (CSU) refractory to antihistamines. This study comprises two parts. In Part 1, participants will be randomized to receive MTPS9579A or placebo. On the basis of positive results from Part 1, a dose-ranging Part 2 may be opened, where participants will be randomized to receive one of four MTPS9579A doses or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CSU refractory to sgH1-AHs at the time of randomization
* Demonstrated ability to comply with the required use of the eDiary for the duration of the study
* For patients on H2 antihistamines or LTRAs for non-CSU indications, treatment at a stable dose for >=2 weeks prior to screening, with no anticipated changes throughout duration of study, including the screening period
* For women of childbearing potential: agreement to remain abstinent or use contraception
* For men: agreement to remain abstinent or use a condom, and agreement to refrain from donating sperm

Exclusion Criteria:

* Previous participation in a clinical trial of MTPS9579A
* Chronic urticaria with known cause or other disease with symptoms of urticaria or angioedema
* Other skin disease associated with chronic itching
* Uncontrolled disease where flares are commonly treated with systemic corticosteroids
* History or evidence of any clinically significant medical condition/disease or abnormalities in laboratory tests that, in the investigator's judgment, preclude the patient's safe participation and completion of the study, or interferes with the conduct and interpretation of the study
* History of anaphylaxis without clearly identifiable avoidable antigen
* History of anaphylaxis to any biologic therapy for any indication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-31 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in the UAS7 | Week 12
  Change from baseline in the Urticaria Activity Score summed over 7 days (UAS7) at Week 12.

SECONDARY OUTCOMES:
Proportion of Participants With Well-Controlled Urticaria | Week 12
  Proportion of participants with well-controlled urticaria (UAS7<=6) at Week 12.
Proportion of Participants Who Achieve Complete Response | Week 12
  Proportion of participants who achieve complete response (UAS7=0) at Week 12.
Percentage of Participants With Adverse Events | Up to approximately 96 weeks
  Percentage of participants with adverse events.
Serum Concentration of MTPS9579A | Through Week 20
Prevalence of Anti-Drug Antibodies (ADAs) | Through Week 20
Incidence of ADAs | Through Week 20

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). Further details on Roche's criteria for eligible studies are available here (https://clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Roche.aspx). For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).